CLINICAL TRIAL: NCT00716495
Title: A Phase I/IIa, Open-label Bridging Safety and Pharmacodynamic Study of a New Formulation of 6 Month Extended Dosing With AGI - 101H Vaccine in the Treatment of Patients With Advanced Melanoma
Brief Title: Safety and Pharmacodynamic Study of a New Formulation, AGI - 101H Vaccine in the Treatment of Advanced Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: problems in funding
Sponsor: AGIRx Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: AGI - 101H/01-2007
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: AGI-101H Vaccine — Each patient will receive one dose of AGI - 101H containing 5 x 107 viable cells, administered s.c. for up to 26 weeks.

SUMMARY:
In this open-label study of patients with advanced melanoma 20 evaluable patients will be recruited.

The drug substance, AGI-101H, is a whole cell, allogeneic melanoma vaccine, representing a mixture (1:1 ratio) of two therapeutic gene modified human melanoma cell lines, referred to as Mich1H6 and Mich2H6, which has been gamma-irradiated to render the cells non-proliferative

Patients will receive treatment for up to 26 weeks. Progression at any time point requiring systemic treatment with, for example with chemotherapy or cytokines will lead to withdrawal of this patient from the study.

The dose chosen is 5 x 107 viable cells/dose.

DETAILED DESCRIPTION:
Total number of patients: 20 evaluable patients will be enrolled in the study.

Dosage: 5 x 107 live cells. No dose modification is planned.

Administration: Subcutaneous (s.c.)

Duration of treatment: Patients will receive treatment for up to 26 weeks. Progression at any time point requiring systemic treatment with, for example with chemotherapy or cytokines will lead to withdrawal of this patient from the study. All surviving patients of this AGITAM trial will be offered the opportunity to transfer to a follow-up treatment protocol with AGI - 101H. In this case treatment may continue every 4 - 8 weeks until progression or death or withdrawal unless such therapy is contraindicated or patient does not wish to continue.

Reference therapy: Not applicable.

Description of medicinal product: The drug substance, AGI-101H, is a whole cell, allogeneic melanoma vaccine, representing a mixture (1:1 ratio) of two therapeutic genemodified human melanoma cell lines, referred to as Mich1H6 and Mich2H6, which has been gamma-irradiated to render the cells non-proliferative. There is no recommended International Non-proprietary (INN) Name for the drug substance.

Methodology: In this open-label study of patients with advanced melanoma, one dose of AGI - 101H vaccine will be administered s.c.. 20 evaluable patients will be recruited. An independent data monitoring committee (DMC) will review all safety data after the first 10 injections and then after another 10 injections (20 injections in total). Up to that second DMC meeting all patients have to stay in the hospital for a 2 hours observation; after the analysis of the 20 vaccinations the DMC will review the safety data and may recommend reverting to normal outpatients setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have given signed informed consent for participation in the study prior to any study-related procedures being performed and not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care
* Age ≥18 years of age and ≤75 years of age
* Histologically confirmed, unresectable stage 3 or 4 measurable (RECIST criteria), cutaneous melanoma or unknown primary with melanoma metastases
* Life expectancy of at least 30 weeks and an ECOG performance status of X 1
* Adequate renal and liver function as defined by serum creatinine and total bilirubin levels no greater than 1.5 times the Investigational Site's upper normal laboratory limits
* Normal clotting
* The patient is willing and able to comply with the protocol for the duration of the study, including 2 hours of follow up observation after the injections (until DMC lifts it after analysis of the first 20 injections) during the course of the trial, examinations and punch biopsies of the vaccination sites 48 hrs post vaccine 1 (week 0) and 8 (week14).

Exclusion Criteria:

* Any previous participation in another trial with the AGI - 101 vaccine
* Ocular or mucosal melanoma
* Pregnant or breast-feeding women, or women of childbearing potential unless effective methods of contraception are used (lack of childbearing potential is met by being post-menopausal, being surgically sterile, practicing contraception with an oral contraceptive or other hormonal therapy [e.g. hormone implants], intra-uterine device, diaphragm with spermicide or condom with spermicide, or being sexually inactive)
* Radiotherapy to target lesions or immunotherapy (including treatment with Interferon or Interleukin-2 and systemic glucocorticosteroids) during the four weeks prior to the start of study treatment.
* Any previous treatment with systemic chemotherapy for advanced melanoma
* Brain metastases
* Major surgery in the four weeks prior to the start of study treatment
* Patients who are poor medical risks due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
* Patients who are known to be serologically positive for Hepatitis B (patients vaccinated against Hepatitis B are accepted), Hepatitis C or HIV
* States causing significant immunosuppression (e.g. organ transplantation or haemodialysis).
* Simultaneous participation in any other study involving investigational drugs or having participated in a study less than 4 weeks prior to start of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The safety profile of AGI-101H | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Gralinska, Study Director — AGIRx (Active Gene Interventions) Ltd
Locations (1):
- WCO (Great Poland Cancer Centre), Poznan, Poland